CLINICAL TRIAL: NCT01596387
Title: Validation of a Pharmacokinetic Pharmacodynamic Model to Administer Propofol in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Ignacio Cortínez F., Profesor Asociado, Departamento de Anestesiología, Pontificia Universidad Catolica de Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-142-Fondecyt-UC-2012
Record Dates: First submitted 2012-05-08; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
Keywords: anaesthetics iv; propofol; pharmacokinetics; pharmacodynamic
MeSH Terms: conditions — Obesity | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Experimental): 20 obese patients(IMC>35 kg m-2) scheduled for laparoscopic bariatric surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — General anesthesia will be induced administering propofol by effect site TCI system using our previously derived model, the target plasma concentration initially will be set at 4 mcg/ml. After loss of consciousness, rocuronium 0.6mg/kg, and remifentanil 0.2mcg/kg/min will be given to facilitate tracheal intubation. After intubation propofol target will be decreased to 3 for 10 minutes and then adapted to the needs of each patient to maintain stable BIS values between 40 and 50. At the end of surgery propofol infusion will be stopped, and patients will be transferred to the recovery unit extubated. Samples of 2.5 ml of arterial blood will be taken at 2, 5 and 10 min after every new target is set. Thereafter samples will be taken at 2, 5, 10, 15, 30, 60, 120 min after stopping drug infusion. Blood samples will be immediately centrifuged and then stored until analysis.

SUMMARY:
The purpose of this study is to validate an integrated pharmacokinetic-pharmacodynamic model to administer propofol in obese patients.

Our hypothesis is that pharmacokinetic and pharmacodynamic changes occur with increasing weight and that mathematical models to administer drugs in obese patients can be developed to accurately predict dose schemes in this population.

DETAILED DESCRIPTION:
Propofol is the most frequently used IV anesthetic today. Propofol TCI is commonly used for induction and maintenance of general anaesthesia in obese and non obese patients. However, current propofol PK models, used in TCI devices, were derived from studies that did not include obese patients. A controversial issue for propofol dose adjustment in this population has been the selection of an adequate size descriptor to scale PK parameters, as drug administration based on total body weight can result in overdose, and conversely, administration based on ideal body weight can result in a sub-therapeutic dose. In a previous study from our group, we developed a PK model capable of characterizing the influence of obesity on propofol disposition. The purpose of this study is to validate this model to administer propofol in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* IMC > 35 kg m-2
* Scheduled for laparoscopic bariatric surgery
* ASA I-II patients
* Between 18 and 60 yr of age.

Exclusion Criteria:

* Patients with allergy to study drugs
* Uncontrolled hypertension
* Heart block greater than first degree
* Take any drug acting in the central nervous system within 24 hrs before surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Validated pharmacokinetic-pharmacodynamic model of Propofol in Obese patients | During the intraoperative period and until 120 min after stopping propofol infusion

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortínez, MD, Principal Investigator — Departamento de Anestesiología, Hospital Clínico Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Cortinez LI, De la Fuente N, Eleveld DJ, Oliveros A, Crovari F, Sepulveda P, Ibacache M, Solari S. Performance of propofol target-controlled infusion models in the obese: pharmacokinetic and pharmacodynamic analysis. Anesth Analg. 2014 Aug;119(2):302-310. doi: 10.1213/ANE.0000000000000317. PMID 24977639